CLINICAL TRIAL: NCT05836896
Title: A Phase I Trial to Establish the Safety and Maximum Tolerated Dose of High-affinity Autologous BCMA-targeting CAR T-cells in Patients With Relapsed and Refractory B-cell Malignancies
Brief Title: A Phase I Trial to Establish the Safety and Maximum Tolerated Dose of High-affinity Autologous BCMA-targeting Chimeric Antigen Receptor (CAR) T-cells in Patients With Relapsed and Refractory B-cell Malignancies
Acronym: CARLOTTA01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUD-BCMACA-078
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms; Relapsed Diffuse Large B-cell Lymphoma (DLBCL); Refractory Diffuse Large B-cell Lymphoma (DLBCL); Multiple Myeloma, Refractory; Multiple Myeloma in Relapse
MeSH Terms: conditions — Neoplasms; Lymphoma, Large B-Cell, Diffuse; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDC-CAR-BCMA001 (Experimental): MDC-CAR-BCMA001 will be administered intravenously in ascending dose levels. This trial will test a total of 4 dose levels in order to identify the MTD and/or recommended phase 2 dose for MDC-CAR-BCMA001.
  Interventions: Genetic: MDC-CAR-BCMA001 (BCMA directed CAR T-cells)

INTERVENTIONS:
Genetic: MDC-CAR-BCMA001 (BCMA directed CAR T-cells) — Single-dose intravenous infusion of MDC-CAR-BCMA001 at the respective dose level following a conditioning chemotherapy

SUMMARY:
The purpose of this phase I study is to determine whether MDC-CAR-BCMA001 (BCMA directed CAR T-cells) is safe and tolerable in the treatment of relapsed and refractory B-cell malignancies

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years
* Written informed consent of the subject
* Able and willing to adhere to the trial protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Either Multiple Myeloma (MM):

  1. relapsed or refractory disease after at least 2 lines of treatment including an Immunomodulatory drug, a proteasome inhibitor and an anti-cluster of differentiation 38 antibody or anti-cluster of differentiation 319 (SLAMF7; Elotuzumab) antibody AND
  2. not eligible for treatment with other regimen available according to local standard of care and known to confer clinical benefit according to the investigator's discretion, prior treatment with other BCMA-targeting immunotherapies (including T-cell engaging antibodies, CAR T-cells and antibody-drug immuno-conjugates) is allowed AND
  3. measurable disease defined by serum M-Protein ≥ 10 g/l OR urine M-Protein ≥ 200 mg/24h OR serum free light chain > 100 mg/l of involved free light chain and abnormal serum free light chain ratio

     OR

     Diffuse large B-cell lymphoma (DLBCL):
  4. Relapsed after or refractory to standard curative therapy (such as R-CHOP) and refractory to at least one course of standard salvage chemotherapy OR
  5. Relapsed within one year after high-dose chemotherapy and autologous stem cell support OR
  6. Relapsed after allogeneic stem-cell transplantation or approved anti-cluster of differentiation 19 CAR T-cell therapies.

     AND (applicable to all DLBCL patients)
  7. Not be eligible for treatment with other regimen available according to local standard of care and known to confer clinical benefit. This includes but is not limited to anti-cluster of differentiation 19 directed CAR T-cell therapies with approved constructs AND (applicable to all DLBCL patients)
  8. Measurable disease according to Lugano criteria
* Adequate organ function defined as:

  1. Neutrophils ≥ 0.5 Gpt/l and Platelets ≥ 50 Gpt/l (unless due to subtotal infiltration of the bone marrow by underlying malignancy)
  2. Lymphocytes ≥ 0.1 Gpt/l
  3. Alaninaminotransferase and Asparataminotransferase ≤ 3.0x Upper limit of normal
  4. Bilirubin ≤ 1.5x Upper limit of normal
  5. Creatinine ≤ 1.5x Upper limit of normal
  6. Adequate cardiac function i.e. left ventricular ejection fraction ≥ 50%, no major valve abnormalities or dyskinesias
* A female of childbearing potential* may be enrolled providing she has a negative pregnancy test at screening and is routinely using a highly effective method of birth control (pearl index of ≤ 1 required) resulting in a low failure rate (e.g. hormonal contraception, intrauterine device, total sexual abstinence or sterilization). Male patients must also prac-tice a highly effective method of birth control and should not father a child at least until 12 months after infusion of CAR T-cells

Exclusion Criteria:

* Any Central nervous system (CNS)-involvement by underlying disease
* History of seizure or cerebrovascular ischemia / hemorrhage within the last 12 months
* History of any autoimmune Central nervous system disease (e.g. multiple sclerosis, amyotrophic lateral sclerosis, optic neuritis)
* Ongoing neurologic conditions that in the opinion of the investigator might increase the risk for neurotoxicity or impair the assessment of CAR-associated neurotoxicity
* Inadequate pulmonary function (i.e. need for continuous oxygen support)
* Patients on hemodialysis
* Any contraindications to Fludarabine and/or Cyclophosphamide as given in the Summary of product characteristics
* Any other active malignancy requiring active treatment or interfering with the assessment of primary or secondary trial endpoints, adjuvant hormonal therapy is allowed
* Positivity for anti-human immunodeficiency virus (HIV) immunoglobulin
* Active or chronic infectious hepatitis B (HBV) and C (HCV) virus unless serology demonstrates clearance of infection (i.e. Polymerase chain reaction undetectable viral load for hepatitis)
* Active infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) or history of SARS-CoV2 infection within the past 3 months or active long coronavirus disease (COVID) syndrome
* Uncontrolled bacterial, viral or fungal infections defined as infections needing in-patient and/or i.v. antimicrobial treatment*
* Active Graft versus Host Disease defined as active symptoms of graft-versus-host disease or ongoing immunosuppressive treatment or prophylaxis within the last 30 days prior to application of MDC-CAR-BCMA001
* Psychologic disorders, drug abuse or any other condition which might significantly impair a patient's ability to comply with the trial protocol
* Patients who are expected to deteriorate during the time needed for manufacturing MDC-CAR-BCMA001 in spite of bridging therapy in the opinion of the investigator including
* Any condition requiring systemic treatment with immunosuppressive drugs (including but not limited to steroids exceeding 20 mg Prednisolone per day)
* Any antineoplastic treatment within 7 days prior to leukapheresis or within 2 weeks or 5 half-lives (whatever is shorter) of the start of lymphodepleting chemotherapy (palliative radiotherapy to lesions not essential for response assessment is allowed without a minimal washout period)
* Any investigational therapy within 4 weeks or 5 half-lives (whatever is shorter) prior to apheresis or the start of lymphodepleting chemotherapy
* History of allergic reactions to any drug or its ingredients / impurities foreseen to be given as part of this trial according to the protocol*
* Receipt of live vaccines within 2 weeks prior to leukapheresis and start of lymphodepleting chemotherapy
* Pregnant or breastfeeding women. Breastfeeding has to be discontinued before onset of and during treatment and should be discontinued for at least 3 months after end of treatment.
* Women of childbearing potential, except women who meet the following criteria:

  1. post-menopausal (12 months natural amenorrhoea or 6 months amenorrhoea with serum Follicle stimulating hormone > 40 U/ml)
  2. postoperative (6 weeks after bilateral ovariectomy with or without hysterectomy)
  3. regular and correct use of a contraceptive method with an Pearl Index < 1% per year
  4. sexual abstinence
  5. Vasectomy of the partner
* Hypersensitivity known from medical history to one of the drugs used or their ingredients or to drugs with a similar chemical structure
* Simultaneous participation in another interventional clinical trial (including within the last 4 weeks before inclusion)
* Addictions or other illnesses that do not allow the person concerned to assess the nature and extent of the clinical trial and its possible consequences
* Indications that the subject is unlikely to adhere to the protocol (e.g., lack of compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of MDC-CAR-BCMA001 | appr. 24 months
  The MTD will be defined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate.
Incidence and severity of adverse events and serious adverse events | appr. 24 months
  graded according to Common Terminology Criteria of Adverse Events V5.0
Incidence and severity of Cytokine release syndrome | appr. 24 months
  Grading of Cytokine release syndrome according to American Society for Transplantation and Cellular Therapy consensus criteria
Incidence and severity of Immune effector cell-associated neurotoxicity syndrome | appr. 24 months
  Grading of Immune effector cell-associated neurotoxicity syndrome according to American Society for Transplantation and Cellular Therapy consensus criteria
Incidence of dose-limiting toxicity (DLT) during DLT-evaluation period and beyond | appr.24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wermke, Prof., Principal Investigator — Technische Universität Dresden (TUD)
Locations (1):
- Technische Universität Dresden, NCT/UCC, Early Clinical Trial Unit, Dresden, Germany